CLINICAL TRIAL: NCT00161915
Title: Prospective Randomized Study on the Efficacy of Endoscopic Injection Therapy With Fibrin Sealant Versus Endoscopic Ligature for Acute Hemostasis and the Prophylaxis of Recurrent Bleeding From Esophageal Varices
Brief Title: Efficacy and Safety of Endoscopic Injection of Fibrin Sealant Versus Endoscopic Ligature for Bleeding Esophageal Varices
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 530001
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-10

CONDITIONS: Esophageal and/or Gastric Varices
Keywords: Liver cirrhosis
MeSH Terms: conditions — Esophageal and Gastric Varices; Liver Cirrhosis | interventions — Fibrin Tissue Adhesive

INTERVENTIONS:
Drug: Fibrin Sealant

SUMMARY:
The purpose of this study was to assess whether endoscopic sclerotherapy with Fibrin Sealant was superior to ligature, with or without Polidocanol, in achieving hemostasis in bleeding esophageal varices and preventing rebleeding. Therapeutic success was defined as survival of the first seven days without clinically significant bleeding.

ELIGIBILITY:
Inclusion Criteria:

Included in the study were patients with proven bleeding from esophageal varices due to liver cirrhosis:

* with a minimum age of 18 years,
* with bleeding symptoms (hematemesis, melena, hematochezia, hypotension, tachycardia) that had lasted not longer than 48 hours prior to hospital admission,
* who were expected to be hospitalized for at least seven days,
* who agreed to participate in the study.

Randomization did not take place if another therapy was medically indicated for any reason.

Exclusion Criteria:

Patients were excluded from the study:

* in whom introduction of an endoscope was not possible for technical reasons,
* who had received an alternative endoscopic treatment to eradicate varices during the last three months (sclerotherapy, ligation),
* who had proven additional fundus bleeding from varices or bleeding from a hypertensive gastropathy,
* who had end stage tumor disease or end stage liver cirrhosis (Child Pugh class C with organ complications, such as hepatonephric syndrome, infected ascites etc.),
* who were pregnant or breast feeding,
* who had a known pulmonary disease combined with restricted lung function or right ventricular failure,
* who had congenital or acquired coagulopathies of non-hepatic origin,
* who were currently participating or had participated in another study during the past 30 days or had already been included in this study once,
* who were treated with drugs to decrease portal vein pressure (somatostatin, somatostatin analogs, terlipressin, glycylpressin, except β-blockers and nitrates),
* who had shown an allergic reaction to thrombin or aprotinin,
* who had a heparin-induced thrombocytopenia Type I or Type II.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zimmer, MD, Principal Investigator — St. Elisabeth Hospital, Wittlich, Germany
Locations (12):
- Germany (12):
  - Helios Klinikum Aue, Aue
  - Krankenhaus Lichtenberg, Berlin
  - Universitätsklinikum Benjamin Franklin, Berlin
  - Krankenhaus Neukölln, Krankenhausbetrieb von Berlin, Berlin
  - Krankenhaus Reinickendorf, Berlin
  - Krankenhaus Zehlendorf, Berlin
  - Klinikum Chemnitz GmbH, Chemnitz
  - Städtisches Klinikum Görlitz, Görlitz
  - Städtisches Klinikum St. Georg, Leipzig
  - Klinikum Ernst von Bergmann, Potsdam
  - St. Josef Krankenhaus, Potsdam
  - St. Elisabeth Krankenhaus, Wittlich